CLINICAL TRIAL: NCT03807141
Title: Evaluation of the Modified Atkins Diet in Children With Epileptic Spasms Refractory to Hormonal Therapy: A Randomized Controlled Trial
Brief Title: Evaluation of the Modified Atkins Diet in Children With Epileptic Spasms
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lady Hardinge Medical College (Other Government)
Responsible Party: Principal Investigator, Suvasini Sharma, Associate Professor, Lady Hardinge Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MADISRCT
Record Dates: First submitted 2019-01-04; First posted 2019-01-16 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Epileptic Spasms
MeSH Terms: conditions — Spasms, Infantile

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet arm (Experimental): Modified Atkins diet will be administered with carbohydrate restriction to 10 grams per day. Proteins will be allowed unrestricted and fats will be actively encouraged.
  The ongoing antiepileptic medication will be continued unchanged
  Interventions: Other: Modified Atkins diet
- Control (No Intervention): The control group will continue their anti-epileptic medication unchanged with no additional dietary input

INTERVENTIONS:
Other: Modified Atkins diet — This is a modified version of the ketogenic diet where-in carbohydrates are restricted without any protein or calorie restriction.
  Arms: Diet arm

SUMMARY:
Epileptic spasms are a difficult to treat epileptic condition in young children. The first line treatment is hormonal treatment, in the form of ACTH or oral steroids, which are effective in 60-70% of children. The condition does not respond well to other anti-epileptic drugs except vigabatrin which is not approved and hence has limited availability and high cost in India. The ketogenic diet, a high fat low carbohydrate diet has been found to be effective in refractory childhood epilepsy especially epileptic spasms. However, the ketogenic diet restricts calories and proteins and required strict weighing of foods. The modified Atkins diet (MAD) is a less restrictive diet which is easier for the parents to prepare and for the children to consume. In this study, it is planned to evaluate the efficacy of the MAD in children with epileptic spasms refractory to hormonal treatment in a randomized controlled trial.

DETAILED DESCRIPTION:
Epileptic spasms comprise an infantile epileptic encephalopathy characterized by hypsarrhythmia on EEG, and frequent neurodevelopmental regression. Unfortunately the treatment of this disorder remains difficult. The first-line options which include hormonal therapy, i.e., adrenocorticotropic hormone (ACTH) or oral corticosteroids, and vigabatrin are effective in 60-70% of the patients. Hormonal therapy is considered the best available treatment. Vigabatrin being expensive and of limited availability is not a feasible option for most patients in our setting. Also, these are associated with significant side effects, and high relapse rates. Newer drugs such as topiramate, zonisamide, and levetiracetam have also been evaluated; however these drugs are less effective than ACTH. The ketogenic diet (KD) is a high fat, low carbohydrate diet. It has been used for treatment of intractable childhood epilepsy. The KD has also been shown in three retrospective studies to be effective for intractable infantile spasms; often after ACTH and vigabatrin have failed. A few previous studies have shown good efficacy of the ketogenic diet on infantile spasms. The traditional ketogenic diet, with 4:1 ratio of fat: carbohydrate + protein has its drawbacks. It restricts calories and fluids, and requires weighing of foods. Protein is generally restricted to 1 g/kg/day, with the majority of remaining calories in the form of fat. This may lead to hypoproteinemia and growth problems. Hospitalization is generally advocated for diet initiation, both for fasting and non-fasting initiation. Side effects of the diet include kidney stones, constipation, acidosis, diminished growth, weight loss, and hyperlipidemia.

The modified Atkins diet is a non-pharmacologic therapy for intractable childhood epilepsy that was designed to be a less restrictive alternative to the traditional ketogenic diet. This diet is started on an outpatient basis without a fast, allows unlimited protein and fat, and does not restrict calories or fluids. Early studies have demonstrated efficacy and safety. Preliminary data have shown efficacy in refractory infantile spasms. Modified Atkins diet may be of special importance in infants, as proteins are not restricted; hence fewer problems with growth are expected. This diet is also ideal for resource-constraint settings with paucity of trained dieticians. Hence this study has been planned to evaluate the efficacy and tolerability of the modified Atkins diet in children with epileptic spasms refractory to hormonal treatment in a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 9 months to 3 years
* Presence of epileptic spasms in clusters in child 9 months to <3years of age, with electroencephalographic evidence of hypsarrhythmia or its variants, persisting, at least one cluster per day, despite treatment with either oral corticosteroids or adrenocorticotrophic hormone (ACTH) and one additional anticonvulsant (valproate/ benzodiazepine/ vigabatrin/ topiramate/ zonisamide/ levetiracetam) for at least 4 weeks.

Exclusion Criteria:

* Children with known or suspected inborn error of metabolism
* Children with renal, pulmonary, cardiac or hepatic dysfunction
* Severe malnutrition (weight for length or weight for height less than -3 Z score as per WHO growth charts)
* Motivational or psychosocial issues in the family which might affect the compliance

Ages: 9 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-01-14 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of children who achieved spasm freedom as per parental reports at 4 weeks, in both the groups | 4 weeks
  The proportion of children who achieve spasm freedom for at least 48 hours as per parental reports at the end of 4 weeks will be evaluated in the both the groups

SECONDARY OUTCOMES:
Proportion of children who achieved >50% reduction of clinical spasm, as per parental reports at 4 weeks, in both the groups. | 4 weeks
  Proportion of children who achieved >50% reduction of clinical spasm, as per parental reports at 4 weeks, in both the groups.
Proportion of children who achieve resolution of hypsarrhythmia on electro encephalogram at 4 weeks in both the groups. | 4 weeks
  Proportion of children who achieve resolution of hypsarrhythmia on electro encephalogram at 4 weeks in both the groups.
Description and proportion of the adverse effects of the diet as per parental reports in the diet group | 4 weeks
  Description and proportion of the adverse effects of the diet as per parental reports in the diet group

CONTACTS AND LOCATIONS:
Locations (1):
- Lady Hardinge Medical College, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharma S, Goel S, Kapoor D, Garg D, Panda I, Elwadhi A, Patra B, Mukherjee SB, Pemde H. Evaluation of the Modified Atkins Diet for the Treatment of Epileptic Spasms Refractory to Hormonal Therapy: A Randomized Controlled Trial. J Child Neurol. 2021 Jul;36(8):686-691. doi: 10.1177/08830738211004747. Epub 2021 Apr 9. PMID 33834913